CLINICAL TRIAL: NCT00573144
Title: Nesiritide Therapy for the Preservation of Left Ventricular Function Post Anterior Myocardial Infarction
Brief Title: Nesiritide Therapy to Preserve Function of the Left Ventricle After Myocardial Infarction
Acronym: Believe II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Horng Chen, Horng Chen, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-002180
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Infusion of 72 hours of saline solution (packaged to match active comparator).
  Interventions: Drug: Placebo
- Nesiritide (Active Comparator): Infusion of 72 hours of IV nesiritide at 0.006 mcg/kg/min.
  Interventions: Drug: Nesiritide

INTERVENTIONS:
Drug: Nesiritide — Infusion of 72 hours of IV nesiritide at 0.006 mcg/kg/min.
  Other Names: Natrecor; BNP
  Arms: Nesiritide
Drug: Placebo — Infusion of 72 hours of saline solution (packaged to match active comparator)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of intravenous human beta natriuretic peptide (BNP, Nesiritide) as compared to placebo to prevent adverse post acute myocardial infarction left ventricular remodeling.

DETAILED DESCRIPTION:
Post acute myocardial infarction (AMI) left ventricular (LV) remodeling begins within hours of the acute event with permanent consequences. Previous studies have demonstrated that LV remodeling is one of the major determinants of long-term survival post AMI. Recent studies have reported that the cardiac natriuretic peptides, atrial natriuretic peptide (ANP) and BNP have direct anti-fibrotic and anti-proliferative effects on the myocardium. More importantly, it has been reported that in the acute phase of AMI, the secretion of the cardiac natriuretic peptides may be insufficient relative to the chronic phase. Therefore, augmentation of the cardiac natriuretic peptide system, such as by exogenous administration of exogenous peptide may prevent post AMI LV remodeling because of the cardioprotective effects. The objective of this study is to to determine the efficacy of IV human BNP (Nesiritide) as compared to placebo to prevent adverse post AMI LV remodeling. This is a randomized double blinded placebo controlled study to determine efficacy of 72 hours of IV BNP at 0.006µg/Kg/min as compared to placebo in patients with anterior ST-elevation myocardial infarction and successful revascularization. The study population will include 60 patients admitted to the Cardiac Care Unit with a first anterior AMI and successful reperfusion therapy (TIMI grade 3 flow) within 24 hours of onset of chest pain documented by coronary angiography.

ELIGIBILITY:
Inclusion criteria:

* Patients with acute ST elevation myocardial infarction with > or = 2 mm ST elevation in one or any combination of anterior leads, with successful revascularization (TIMI grade 3 flow) of the lesion within 24 hours of symptoms and consented within 24 hours of procedure.

Exclusion criteria:

* Cardiogenic shock or hypotension, Systolic BP< 90 mmHg or overt Congestive Heart Failure (CHF)
* Previous history of MI (Myocardial Infarction)
* Previous ECG suggesting previous MI
* Known Ejection Fraction (EF) < 30%
* Atrial fibrillation
* Previously known significant valvular disease (Grade III, IV), cardiomyopathy and congenital heart disease.
* Hemoglobin <10 mg/dL
* Pregnant women/nursing mothers
* Participants still menstruating and have not been surgically sterilized must have a negative pregnancy test prior to participating in this study.
* Unable to undergo cardiac MRI (Magnetic Resonance Imaging).
* Contraindications to MRI include pacemaker or defibrillator, pregnant women, atrial fibrillation or other arrhythmia, cerebral aneurysm clips or severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-09; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H. Chen, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonvilee, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Hubers SA, Schirger JA, Sangaralingham SJ, Chen Y, Burnett JC Jr, Hodge D, Chen HH. B-type natriuretic peptide and cardiac remodelling after myocardial infarction: a randomised trial. Heart. 2021 Mar;107(5):396-402. doi: 10.1136/heartjnl-2020-317182. Epub 2020 Aug 3. PMID 32747497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Mayo Clinic Cardiac Care Units in Rochester, Minnesota and Jacksonville, Florida.
Pre-assignment Details: One subject withdrew consent before randomization.
Period: Overall Study
Arm/Group | Placebo | Nesiritide
Started | 30 | 28
Completed | 28 | 25
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline values are reported for subjects completing the study (28 in placebo group and 25 in nesiritide group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nesiritide | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.85 (11.12) | 60.4 (11.15) | 58.0 (11.26)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 17 | 39
  >=65 years | 6 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 25 | 22 | 47
Region of Enrollment [Number; unit: participants]
  United States | 28 | 25 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End-Systolic Volume Index
Description: Change in Left Ventricular end-systolic volume index as determined by Multiple Gated Acquisition (MUGA) scan from baseline to 30 days. The MUGA scan is a noninvasive tool for assessing the function of the heart. The MUGA scan produces a moving image of the beating heart, and from this image several important features can be determined about the health of the cardiac ventricles (the heart's major pumping chambers). End-systolic volume (ESV) is the volume of blood in a ventricle at the end of contraction, or systole, and the beginning of filling, or diastole. ESV is the lowest volume of blood in the ventricle at any point in the cardiac cycle and can be used clinically as a measurement of the adequacy of cardiac emptying, related to systolic function.
Time Frame: baseline, 30 days
Measure: Mean (Standard Deviation); unit: mL of blood/meter^2 body surface area
Arm/Group | Placebo | Nesiritide
Number analyzed (Participants) | 28 | 25
mL of blood/meter^2 body surface area | -2.1 (58) | -4.6 (31)
Statistical Analysis 1: Comparison: Placebo vs Nesiritide; Test type: Superiority or Other; p = 0.97, t-test, 2 sided

2. Secondary Outcome: Change in Left Ventricular End-Systolic Diastolic Volume Index
Description: Change in Left Ventricular end-systolic diastolic volume index determined by Multiple Gated Acquisition (MUGA) scan from baseline to 30 days. The MUGA scan is a noninvasive tool for assessing the function of the heart. The MUGA scan produces a moving image of the beating heart, and from this image several important features can be determined about the health of the cardiac ventricles (the heart's major pumping chambers). End-systolic volume (ESV) is the volume of blood in a ventricle at the end of contraction, or systole, and the beginning of filling, or diastole. ESV is the lowest volume of blood in the ventricle at any point in the cardiac cycle and can be used clinically as a measurement of the adequacy of cardiac emptying, related to systolic function.
Time Frame: baseline, 30 days
Measure: Mean (Standard Deviation); unit: mL blood/meter^2 body surface area
Arm/Group | Placebo | Nesiritide
Number analyzed (Participants) | 28 | 25
mL blood/meter^2 body surface area | 4.4 (88) | 9.7 (51)
Statistical Analysis 1: Comparison: Placebo vs Nesiritide; Test type: Superiority or Other; p = 0.35, t-test, 2 sided

3. Secondary Outcome: Myocardial Infarct Size at 30 Days
Description: Myocardial infarction or acute myocardial infarction (AMI) is the medical term for an event commonly known as a heart attack. Myocardial (heart muscle) infarction is tissue death (also known as necrosis) caused by a local lack of oxygen, due to an obstruction of the tissue's blood supply. The resulting heart tissue lesion is referred to as an infarct. A larger size or area of infarct indicates a greater amount of heart tissue death. Myocardial infarct size was measured using a cardiac Magnetic Resonance Imaging (MRI) scan at 30 days and is the mass of the infarcted tissue divided by the mass of the left ventricle times 100%.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: percentage of total cardiac tissue mass
Arm/Group | Placebo | Nesiritide
Number analyzed (Participants) | 28 | 25
percentage of total cardiac tissue mass | 17 (14) | 12 (9)
Statistical Analysis 1: Comparison: Placebo vs Nesiritide; Test type: Superiority or Other; p = 0.26, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Placebo | Nesiritide
Serious Adverse Events (participants affected / at risk) | 5/28 | 1/25
Other Adverse Events (participants affected / at risk) | 13/28 | 13/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Nesiritide (N=25)
Left ventricle aneurysm or thrombus (Cardiac disorders) | 2 (2) | 1 (1)
Hospital readmission for chest pain (Cardiac disorders) | 2 (2) | 0 (0)
Hospital readmission for other reasons (not chest pain) (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Nesiritide (N=25)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Post coronary angiogram related complications (Cardiac disorders) | 4 (4) | 3 (3)
Subsequent coronary angiogram with no intervention (Cardiac disorders) | 2 (2) | 1 (1)
Subsequent coronary angiogram with intervention other than LAD (Cardiac disorders) | 3 (3) | 1 (1)
Persistent ECG ST changes (Cardiac disorders) | 0 (0) | 1 (1)
Recurrent chest pain (Cardiac disorders) | 1 (1) | 1 (1)
Vasovagal spell (Cardiac disorders) | 1 (1) | 0 (0)
MRI dye allergy (General disorders) | 1 (1) | 0 (0)
Asthma flare (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 2 (2) | 0 (0)
First episode of hypotension (asymptomatic) (Cardiac disorders) | 13 (13) | 13 (13)
First episode of hypotension (symptomatic) (Cardiac disorders) | 0 (0) | 2 (2)
Second episode of hypotension (asymptomatic) (Cardiac disorders) | 7 (7) | 10 (10)
Second episode of hypotension (symptomatic) (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No